CLINICAL TRIAL: NCT02070198
Title: Long Acting FSH Plus GnRH Antagonist Versus Daily FSH Plus GnRH Antagonist Versus Short Agonist Regimens in Poor Responder Patients Undergoing IVF: a Randomized Study.
Brief Title: Long Acting FSH Plus Antagonist Versus Daily FSH Plus Antagonist Versus Short Agonist Protocol in Poor Responders Undergoing IVF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bioroma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRM001
Record Dates: First submitted 2014-02-20; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Female Infertility; Poor Responder
Keywords: Poor responders, IVF, GnRH agonist, GnRH antagonist, recombinant FSH
MeSH Terms: conditions — Infertility, Female | interventions — Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Long acting FSH and GnrH antagonist (Experimental): Woman in long acting FSH and GnRH antagonist arm receive an initial dose of 150 mcg Corifollitropin alfa on second day of the menstrual cycle followed by a fixed daily dose of 0.25 mg of GnRH antagonist on day 7 of the cycle onwards. On the ninth day of the cycle, a daily fixed dose of 300 IU of recombinant FSH will be administered until the day of ovulation triggering.
  Interventions: Drug: Long acting FSH and GnRH antagonist
- daily FSH and GnRH antagonist (Experimental): Woman in daily FSH and GnRH antagonist arm receive a fixed dose of 300 IU of recombinantFSH starting 3 day of the menstrual cycle followed by a fixed daily dose of 0.25 mg of GnRH antagonist on day 7 of the cycle onwards until the day of ovulation triggering.
  Interventions: Drug: Daily FSH and GnRH antagonist
- Triptorelin and recombinant FSH (Experimental): Women in triptorelin and recombinant FSH arm receive a fixed dose of 0.05 mg of triprorelin from the 1 day of the menstrual cycle followed by a fixed dose of 300 IU of recombinant FSH starting 3 day until the day of HCG administration.
  Interventions: Drug: Triptorelin and recombinant FSH

INTERVENTIONS:
Drug: Long acting FSH and GnRH antagonist — Woman in long acting FSH and GnRH antagonist arm receive an initial dose of 150 mcg Corifollitropin alfa on second day of the menstrual cycle followed by a fixed daily dose of 0.25 mg of GnRH antagonist on day 7 of the cycle onwards. On the ninth day of the cycle, a daily fixed dose of 300 IU of recombinant FSH will be administered until the day of ovulation triggering.
  Arms: Long acting FSH and GnrH antagonist
Drug: Daily FSH and GnRH antagonist — Woman in daily FSH and GnRH antagonist arm receive a fixed dose of 300 IU of recombinantFSH starting 3 day of the menstrual cycle followed by a fixed daily dose of 0.25 mg of GnRH antagonist on day 7 of the cycle onwards until the day of ovulation triggering.
  Arms: daily FSH and GnRH antagonist
Drug: Triptorelin and recombinant FSH — Women in Triptorelin and recombinant FSH arm receive a fixed dose of 0.05 mg of Triprorelin from the 1 day of the menstrual cycle followed by a fixed dose of 300 IU of recombinant FSH starting 3 day untill the day of HCG administration.
  Arms: Triptorelin and recombinant FSH

SUMMARY:
Despite the progression in assisted reproductive technology (ART), poor ovarian response to controlled ovarian stimulation remains a challenge for clinicians and a source of distress for patients. Multiple strategies have been tried to overcome these obstacles. The increase of the gonadotropin administration have been associated with a very low pregnancy rate. The introduction of GnRH agonist protocol, which takes advantage of the initial rise in endogenous gonadotropins that follows the agonist administration in the early follicular phase and subsequently prevents a premature LH surge, with fewer cycle cancellations, have improved cycle parameters and increased pregnancy rate. Recently, GnRH antagonists were introduced in ART treatment. They are effective in preventing a premature LH surge and allow for a more natural recruitment of follicles in the follicular phase in a non suppressed ovary. However, the randomized studies comparing the efficacy of these two regimens reported conflicting and nonsignificant results. Moreover, more recently adjuvant therapies for COH such as growth hormone therapy or pyridostigmine, oral L-arginine, and transdermal testosterone failed to improve IVF outcomes. Recently, the new treatment option with corifollitropin alfa, able to keep the circulating FSH level above the threshold necessary to support multi-follicular growth for an entire week, in a GnRH antagonist protocol seems to have a potential beneficial effect in poor responders.

The aim of this study is to compare long-acting FSH/GnRH antagonist with daily FSH/GnRH antagonist with short GnRH agonist protocol on IVF outcome in poor responder patients .

ELIGIBILITY:
Inclusion Criteria:

* women with at least two of the following criteria: I) age > 40 years old; II) basal follicular stimulation hormone (FSH) > 12 mIU/ml; III) three or fewer oocytes retrieved in the previous IVF cycle; IV) low estradiol levels on the day of human chorionic gonadotropin (hCG) administration (< 1500 pmol/ml).

Exclusion Criteria:

* body mass index > 30
* biochemical and ultrasound evidence of polycystic ovary syndrome
* stage III-IV endometriosis
* inflammatory or autoimmune disorders
* metabolic disease
* infertility medications (gonadotropins, clomiphene citrate) within the past two months

Ages: 25 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | Time Frame: until 12th gestational week

SECONDARY OUTCOMES:
Implantation rate | Time Frame: until 12th gestational week

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Schimberni, MD, Principal Investigator — Bioroma
Locations (1):
- Bioroma, Rome, Italy, Italy